CLINICAL TRIAL: NCT01170832
Title: Cardiac Autonomic Neuropathy and Myocardial Dysfunction in Type 1 Diabetes
Brief Title: To Evaluate if Wide Blood Sugar Fluctuations Lead to Injury of Heart Function and Heart Nerves
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Professor of Internal Medicine/MEND, University of Michigan
Other Study IDs: HUM 00036408
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect approximately 15 ml of whole blood for DNA sampling and storage.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This proposal will test if, in patients with type 1 diabetes, wide blood glucose fluctuations lead to the injury to heart nerves , called cardiac autonomic neuropathy (CAN), and to impaired heart contractile (pumping) function and heart failure. It will also evaluate the natural history of heart failure and enhanced cardiac risk in patients with type 1 diabetes in the current standard of diabetes care.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Male or female between the ages 18-65, with type 1 diabetes of 5-10 years duration who are free of complications and age-and-sex-matched healthy control volunteers.
* Hemoglobin A1c greater than 7 %. (For Type 1 diabetics)
* If you are a woman of childbearing potential you must agree to use an acceptable birth control method throughout the duration of the study. The methods of birth control that you can use are: Oral contraceptives (birth control pill), IUD or a barrier method (e.g. diaphragm or condom with spermicide).
* You should have no history of any cardiovascular disease including any form of coronary artery disease, congestive heart failure, known arrhythmias (irregular heart beats), valvular disease or high blood pressure.
* If you have any pacemaker or ICD, if you have any metallic foreign body such as surgical implants or clips or foreign bodies in the eye or orbits, wearing medication patches containing foil, or any other metal in the body or if you are claustrophobic you cannot participate in this study.
* You should be free of any diabetic complications (e.g. nephropathy or kidney damage, retinopathy or eye damage), have no history of previous kidney, pancreas or cardiac transplantation, any other severe chronic illness that has neuropathy (numbness, burning or tingling) and/or neurologic disease as a recognized complication (e.g. Parkinson's disease, epilepsy), or any other serious medical conditions that may shorten life span (e.g. disabling stroke, Chronic Obstructive Pulmonary Disease).
* You should be free of any malignancy other than basal cell skin cancer.
* No history of alcohol abuse.
* You should not use any agents or drugs that interfere with the imaging techniques described below.
* You must be able to cooperate with the test protocols that are described below and be willing to sign this consent form.

Inclusion for Control group:

* BMI <30
* If female, must not be pregnant or nursing
* Normal blood pressure
* Normal labs-(glucose and lipids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetics who have been diagnosed between 5-10 years and do not have any complications that are associated with Diabetes
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2010-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Heart rate (HR) Variability Studies | Three years
  Evaluation of heart rate variability and 24 hour blood pressure monitoring: electrocardiogram (ECG) and blood pressure will be recorded while resting in a lying down position and during certain controlled procedures that include deep breathing and other clinical maneuvers such as standing up and exhaling deeply.

SECONDARY OUTCOMES:
Positron Emission Tomography (PET) scan | Test to be completed at baseline and end of study (3yrs)
  Subjects will have a heart positron emission tomography (PET) scan, using a radioisotope called [11C] hydroxyl-ephedrine (HED). This type of heart PET scan allows mapping the heart nerves. You will also have another scan with a radioisotope called [11C]-acetate which will help us measure the metabolism of your heart and how efficiently it contracts.

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, MD, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- University Of Michigan, Ann Arbor, Michigan, United States